CLINICAL TRIAL: NCT01088334
Title: Trousseau Studie, Mortaliteit Door Maligniteit Bij patiënten Met Idiopatische Veneuze Tromboembolie
Brief Title: Mortality Due to Malignancy in Patients With Idiopathic Venous Thromboembolism
Acronym: Trousseau
Status: Terminated | Type: Observational
Why Stopped: Terminated because of futility to continue, after planned interim analysis.
Sponsor: Slotervaart Hospital (Other)
Responsible Party: Dr. JMMB Otten, pi, Slotervaart hospital
Other Study IDs: Trousseau studie
Record Dates: First submitted 2010-02-25; First posted 2010-03-17 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-03

CONDITIONS: Venous Thromboembolism; Malignancy
Keywords: Idiopathic venous thromboembolism; Malignancy; screening
MeSH Terms: conditions — Venous Thromboembolism; Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- IVTE, follow-up: no malignancy at basal screening, no extensive screening
- IVTE, screening: No malignancy at basal screening, screening by means of CT-Chest/abdomen and mammography in women
  Interventions: Other: screening

INTERVENTIONS:
Other: screening — CT-Chest/abdomen and mammography in women
  Groups: IVTE, screening

SUMMARY:
Background

Patients with an idiopathic venous thromboembolism (IVTE) appear to have a risk of approximately 10% for symptomatic malignancy within 3 years after the IVTE. It is not clear if extensive screening for malignant disease leads to survival benefit in patients with an IVTE.

The SOMIT study learned that it is feasible to screen patients with an IVTE for malignancy and screening by means of a computer tomography (CT) of the chest and abdomen plus a mammography in women had the potential to be most cost-effective. The SOMIT study could not show a survival benefit due to the design of the study.

Primary objective: cancer related mortality

Methods:

The Trousseau study has been designed as a multicenter, prospective concurrently controlled cohort study.

Inclusion criteria:

1. Proven first symptomatic deep venous thromboembolic event;
2. Without: known risk factor for venous thromboembolism.

Exclusion criteria:

1. Proven deep venous thromboembolic event in the medical history, age under 40 years;
2. Patients without signs of malignancy after routine investigations (medical history, physical examination, laboratory investigations and chest X-ray) were included. Depending on the standard care in the hospital of interest, one group of patients has been screened by means of CT-chest and abdomen plus mammography, the other group had no additional investigations. Follow-up was aimed to be 3 years in both groups (at 3, 6, 12, 24 and 36 months after the thromboembolic event).

Data like mortality rate, morbidity due to screening procedures, additional investigations, number of cancer patients detected by the extensive screening, number of cancer patients three years after the IVTE, number and kind of investigations performed and information about cancer treatment and hospitalization was collected. If this information indicate a survival benefit these data enable us to perform a cost-effectiveness analysis.

Endpoint: Mortality.

Statistics:

Based on the prevalence of occult malignancy in VTE patients, the nature and stage of malignancies, the expected mortality, the anticipated detection of cancers and the early treatment related decrease in mortality we needed, in order to detect a true difference of this size with a 80 percent power and a two-tailed certainty of five percent, 750 patients for each group. Therefore, a total of 1500 patients is required for this study.

DETAILED DESCRIPTION:
Study design:

Although a randomized design is ideal for most studies we preferred a multicenter, prospective concurrently controlled cohort study design for our study. This is based on the experiences with the SOMIT study, in which two of the members of the executive committee (MH Prins, JMMB Otten) were involved.

The SOMIT study originally was supposed to have been conducted in eight countries. Medical ethical committees in most countries however considered it unethical to conduct this randomized study. Either because of the fact that the study contained a control arm, or because the screening arm (and thus the study itself) was considered to be unethical.

Patients as well as physicians found it difficult to let fate decide whether or not a patient would be screened for cancer, even though it was not clear if screening was life-saving. Moreover, during the SOMIT study, physicians noticed that patients with IVTE had their cancer detected early if they were in the screening group. This made it even more difficult to withhold additional screening procedures in patients in the routine group.

Many physicians themselves showed a strong preference for one of the arms of the study. Therefore they did not include as many patients as they could.

With a prospective cohort design we expect to avoid these problems. Per hospital that participates in the Trousseau study the physicians in that hospital will treat the patients according to the local preference for screening or no screening. All hospitals are matched regarding their population as much as possible.

Statistics:

The prevalence of occult cancer at the time of the thrombotic episode in patients with IVTE can be estimated to be 10%. Based on the nature and stage of malignancies, it is expected that half of these patients with occult malignant disease will die during the 3 years of follow-up, resulting in a cancer-related mortality of 5%. In addition, in approximately half of the patients with malignant disease who survived for 3 years, residual or recurrent cancer will be present. Therefore, cancer-related mortality or residual or recurrent cancer will be present in 75% of the patients with occult malignant disease at presentation, i.e., in 7-8% of the patients of the study cohort. We anticipate that approximately 80% of the occult malignancies will be detected by extensive screening and that early treatment will result in a 50% to 75% reduction of the 3-year incidence of cancer-related mortality or residual or recurrent malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Proven first symptomatic deep venous thromboembolic event;
* No known malignancy
* Without: trauma of the legs, surgery within the last 2 months, immobilization within the last 2 months, thrombocytosis (> 1000 x 109), clinical severe dehydration, deficiency of anti-thrombin III, protein C/S, Factor V Leiden mutation , Prothrombine mutation or circulating lupus anticoagulants, pregnancy or post-partum period
* No indication for malignancy at routine investigations(medical history, physical examination, routine blood tests and chest X-ray)

Exclusion Criteria:

* Proven deep venous thromboembolic event in the medical history
* age under 40 years;

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with IVTE diagnosed in academical centres and teaching hospitals in the Netherlands
Sampling Method: Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2002-12; Primary Completion 2008-05 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Mortality | at 3, 6, 12, 24, 36 months after inclusion and at the end of study
  The responsible physician inform the investigators when a patient has died. The national registrar was checked at the end of the study for all patients

SECONDARY OUTCOMES:
Residual objectified malignancy | at 3, 6, 12, 24, 36 months after inclusion
  The responsible physician documented all investigations performed. The malignancy have to be objectified. At the end of the study all living patients were contacted for medical status.
Recurrent objectified malignancy | at 3, 6, 12, 24, 36 after inclusion.
  The responsible physician documented all investigations performed. The malignancy have to be objectified. At the end of the study all living patients were contacted for medical status.
Malignancy detected by extensive screening, without alarm signs in routine examinations | at 3 months after inclusion
  The responsible physician documented all investigations performed and documented in standardized manner the routine tests (medical history, physical examination, lab tests and Chest X-ray. The malignancy have to be objectified inconnection with and due to screening tests and eventually further investigations.
Costs of screening, of additional tests after screening | at end of study.
  All costs of routine tests (consult of phycisians, lab tests, X-Chest) are known and documented, as are the costs of the screening tests and, if performed the costs of further evaluation in case of additional tests, admitions etc..
Medical complications of screening tests | at 3 + 6 months and end of study
  The screening tests had no risk of damage other than radiation. The results of these tests however could urge for invasive tests that could potentially harm patients. Therefore the harm done by screening tests or the resulting tests were documented.

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Martin MB Otten, MD PhD, Principal Investigator — Slotervaart hospital and Academic Medical Center; Harry R Büller, Md PhD, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Martin H Prins, MD PhD, Study Chair — Maastricht Universitair Medisch Centrum; Frederiek F v. Doormaal, MD PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Wim Terpstra, MD PhD, Study Chair — Onze Lieve Vrouwe Gasthuis; René vd Griend, MD PhD, Study Chair — Diakonessenhuis, Utrecht; Marten Nijziel, MD PhD, Study Chair — Maxima Medical Center; Marcel A vd Ree, MD PhD, Study Chair — Diakonessenhuis Zeist; Jacob C Dutilh, MD, Study Chair — Meander Medisch Centrum; A t. Cate-Hoek, MD PhD, Study Chair — Maastricht Universitair Medisch Centrum; Simone M. vd Heiligenberg, MD, Study Chair — Dijklander Ziekenhuis; Jan vd Meer, MD PhD, Study Chair — University Medical Center Groningen
Locations (10):
- Netherlands (10):
  - Meander Medisch Centrum, Amersfoort
  - Slotervaarthospital, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academic Medical Center, Amsterdam
  - Maxima Medisch Centrum, Eindhoven
  - Academisch Ziekenhuis Groningen, Groningen
  - Westfries Gasthuis, Hoorn
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Diakonessenhuis Utrecht, Utrecht
  - Diakonessenhuis Zeist, Zeist

REFERENCES:
- [Background] Bastounis EA, Karayiannakis AJ, Makri GG, Alexiou D, Papalambros EL. The incidence of occult cancer in patients with deep venous thrombosis: a prospective study. J Intern Med. 1996 Feb;239(2):153-6. doi: 10.1046/j.1365-2796.1996.426000.x. PMID 8568483
- [Background] Carson JL, Kelley MA, Duff A, Weg JG, Fulkerson WJ, Palevsky HI, Schwartz JS, Thompson BT, Popovich J Jr, Hobbins TE, et al. The clinical course of pulmonary embolism. N Engl J Med. 1992 May 7;326(19):1240-5. doi: 10.1056/NEJM199205073261902. PMID 1560799
- [Background] Griffin MR, Stanson AW, Brown ML, Hauser MF, O'Fallon WM, Anderson HM, Kazmier FJ, Melton LJ 3rd. Deep venous thrombosis and pulmonary embolism. Risk of subsequent malignant neoplasms. Arch Intern Med. 1987 Nov;147(11):1907-11. PMID 3675090
- [Background] Goldberg RJ, Seneff M, Gore JM, Anderson FA Jr, Greene HL, Wheeler HB, Dalen JE. Occult malignant neoplasm in patients with deep venous thrombosis. Arch Intern Med. 1987 Feb;147(2):251-3. PMID 3813741
- [Background] Monreal M, Salvador R, Soriano V, Sabria M. Cancer and deep venous thrombosis. Arch Intern Med. 1988 Feb;148(2):485. No abstract available. PMID 3341848
- [Background] Gore JM, Appelbaum JS, Greene HL, Dexter L, Dalen JE. Occult cancer in patients with acute pulmonary embolism. Ann Intern Med. 1982 May;96(5):556-60. doi: 10.7326/0003-4819-96-5-556. PMID 7073147
- [Background] Monreal M, Lafoz E, Casals A, Inaraja L, Montserrat E, Callejas JM, Martorell A. Occult cancer in patients with deep venous thrombosis. A systematic approach. Cancer. 1991 Jan 15;67(2):541-5. doi: 10.1002/1097-0142(19910115)67:23.0.co;2-j. PMID 1985747
- [Background] Aderka D, Brown A, Zelikovski A, Pinkhas J. Idiopathic deep vein thrombosis in an apparently healthy patient as a premonitory sign of occult cancer. Cancer. 1986 May 1;57(9):1846-9. doi: 10.1002/1097-0142(19860501)57:93.0.co;2-3. PMID 3955523
- [Background] Hettiarachchi RJ, Lok J, Prins MH, Buller HR, Prandoni P. Undiagnosed malignancy in patients with deep vein thrombosis: incidence, risk indicators, and diagnosis. Cancer. 1998 Jul 1;83(1):180-5. doi: 10.1002/(sici)1097-0142(19980701)83:13.0.co;2-s. PMID 9655309
- [Background] Monreal M, Fernandez-Llamazares J, Perandreu J, Urrutia A, Sahuquillo JC, Contel E. Occult cancer in patients with venous thromboembolism: which patients, which cancers. Thromb Haemost. 1997 Nov;78(5):1316-8. PMID 9408011
- [Background] Rajan R, Levine M, Gent M, Hirsh J, Geerts W, Skingley P, Julian J. The occurrence of subsequent malignancy in patients presenting with deep vein thrombosis: results from a historical cohort study. Thromb Haemost. 1998 Jan;79(1):19-22. PMID 9459315
- [Background] Prins MH, Hettiarachchi RJ, Lensing AW, Hirsh J. Newly diagnosed malignancy in patients with venous thromboembolism. Search or wait and see? Thromb Haemost. 1997 Jul;78(1):121-5. PMID 9198140
- [Background] O'Connor NT, Cederholm-Williams SA, Fletcher EW, Allington M, Sharp AA. Significance of idiopathic deep venous thrombosis. Postgrad Med J. 1984 Apr;60(702):275-7. doi: 10.1136/pgmj.60.702.275. PMID 6539470
- [Background] Prandoni P, Lensing AW, Buller HR, Cogo A, Prins MH, Cattelan AM, Cuppini S, Noventa F, ten Cate JW. Deep-vein thrombosis and the incidence of subsequent symptomatic cancer. N Engl J Med. 1992 Oct 15;327(16):1128-33. doi: 10.1056/NEJM199210153271604. PMID 1528208
- [Background] Lensing AW, Prandoni P, Brandjes D, Huisman PM, Vigo M, Tomasella G, Krekt J, Wouter Ten Cate J, Huisman MV, Buller HR. Detection of deep-vein thrombosis by real-time B-mode ultrasonography. N Engl J Med. 1989 Feb 9;320(6):342-5. doi: 10.1056/NEJM198902093200602. PMID 2643771
- [Background] Rance A, Emmerich J, Guedj C, Fiessinger JN. Occult cancer in patients with bilateral deep-vein thrombosis. Lancet. 1997 Nov 15;350(9089):1448-9. doi: 10.1016/S0140-6736(05)64210-9. No abstract available. PMID 9371175
- [Background] Sannella NA, O'Connor DJ Jr. "Idiopathic" deep venous thrombosis: the value of routine abdominal and pelvic computed tomographic scanning. Ann Vasc Surg. 1991 May;5(3):218-22. doi: 10.1007/BF02329376. PMID 2064913
- [Background] Cornuz J, Pearson SD, Creager MA, Cook EF, Goldman L. Importance of findings on the initial evaluation for cancer in patients with symptomatic idiopathic deep venous thrombosis. Ann Intern Med. 1996 Nov 15;125(10):785-93. doi: 10.7326/0003-4819-125-10-199611150-00001. PMID 8928984
- [Background] Carrier M, Le Gal G, Wells PS, Fergusson D, Ramsay T, Rodger MA. Systematic review: the Trousseau syndrome revisited: should we screen extensively for cancer in patients with venous thromboembolism? Ann Intern Med. 2008 Sep 2;149(5):323-33. doi: 10.7326/0003-4819-149-5-200809020-00007. PMID 18765702
- [Background] Buller HR, Davidson BL, Decousus H, Gallus A, Gent M, Piovella F, Prins MH, Raskob G, Segers AE, Cariou R, Leeuwenkamp O, Lensing AW; Matisse Investigators. Fondaparinux or enoxaparin for the initial treatment of symptomatic deep venous thrombosis: a randomized trial. Ann Intern Med. 2004 Jun 1;140(11):867-73. doi: 10.7326/0003-4819-140-11-200406010-00007. PMID 15172900
- [Background] Girolami A, Prandoni P, Zanon E, Bagatella P, Girolami B. Venous thromboses of upper limbs are more frequently associated with occult cancer as compared with those of lower limbs. Blood Coagul Fibrinolysis. 1999 Dec;10(8):455-7. doi: 10.1097/00001721-199912000-00001. PMID 10636455
- [Background] Ahmed Z, Mohyuddin Z. Deep vein thrombosis as a predictor of cancer. Angiology. 1996 Mar;47(3):261-5. doi: 10.1177/000331979604700307. PMID 8638869
- [Background] Subira M, Mateo J, Souto JC, Altes A, Fontcuberta J. Lack of association between venous thrombosis and subsequent malignancy in a retrospective cohort study in young patients. Am J Hematol. 1999 Mar;60(3):181-4. doi: 10.1002/(sici)1096-8652(199903)60:33.0.co;2-4. PMID 10072107
- [Background] Biello DR, Mattar AG, McKnight RC, Siegel BA. Ventilation-perfusion studies in suspected pulmonary embolism. AJR Am J Roentgenol. 1979 Dec;133(6):1033-7. doi: 10.2214/ajr.133.6.1033. PMID 116491
- [Background] Dalen JE, Brooks HL, Johnson LW, Meister SG, Szucs MM Jr, Dexter L. Pulmonary angiography in acute pulmonary embolism: indications, techniques, and results in 367 patients. Am Heart J. 1971 Feb;81(2):175-85. doi: 10.1016/0002-8703(71)90128-1. No abstract available. PMID 5539544
- [Background] Hull RD, Hirsh J, Carter CJ, Raskob GE, Gill GJ, Jay RM, Leclerc JR, David M, Coates G. Diagnostic value of ventilation-perfusion lung scanning in patients with suspected pulmonary embolism. Chest. 1985 Dec;88(6):819-28. doi: 10.1378/chest.88.6.819. PMID 4064769
- [Background] PIOPED Investigators. Value of the ventilation/perfusion scan in acute pulmonary embolism. Results of the prospective investigation of pulmonary embolism diagnosis (PIOPED). JAMA. 1990 May 23-30;263(20):2753-9. doi: 10.1001/jama.1990.03440200057023. PMID 2332918
- [Background] Otten HM, Prins MH. A number needed to screen and cost-effectiveness analysis of the SOMIT-data. Haemostasis. 2001;31 Suppl 1:40-2. No abstract available. PMID 11990474
- [Background] Piccioli A, Prandoni P. Screening for occult cancer in patients with idiopathic venous thromboembolism: yes. J Thromb Haemost. 2003 Nov;1(11):2271-2. doi: 10.1046/j.1538-7836.2003.00505.x. No abstract available. PMID 14629455
- [Background] Lee AY. Screening for occult cancer in patients with idiopathic venous thromboembolism: no. J Thromb Haemost. 2003 Nov;1(11):2273-4. doi: 10.1046/j.1538-7836.2003.00490.x. No abstract available. PMID 14629456
- [Background] Monreal M, Lensing AW, Prins MH, Bonet M, Fernandez-Llamazares J, Muchart J, Prandoni P, Jimenez JA. Screening for occult cancer in patients with acute deep vein thrombosis or pulmonary embolism. J Thromb Haemost. 2004 Jun;2(6):876-81. doi: 10.1111/j.1538-7836.2004.00721.x. PMID 15140120
- [Background] Piccioli A, Lensing AW, Prins MH, Falanga A, Scannapieco GL, Ieran M, Cigolini M, Ambrosio GB, Monreal M, Girolami A, Prandoni P; SOMIT Investigators Group. Extensive screening for occult malignant disease in idiopathic venous thromboembolism: a prospective randomized clinical trial. J Thromb Haemost. 2004 Jun;2(6):884-9. doi: 10.1111/j.1538-7836.2004.00720.x. PMID 15140122
- [Background] DI Nisio M, Otten HM, Piccioli A, Lensing AW, Prandoni P, Buller HR, Prins MH. Decision analysis for cancer screening in idiopathic venous thromboembolism. J Thromb Haemost. 2005 Nov;3(11):2391-6. doi: 10.1111/j.1538-7836.2005.01606.x. PMID 16241936
- [Background] Nordstrom M, Lindblad B, Anderson H, Bergqvist D, Kjellstrom T. Deep venous thrombosis and occult malignancy: an epidemiological study. BMJ. 1994 Apr 2;308(6933):891-4. doi: 10.1136/bmj.308.6933.891. PMID 8173368
- [Background] Sorensen HT, Mellemkjaer L, Steffensen FH, Olsen JH, Nielsen GL. The risk of a diagnosis of cancer after primary deep venous thrombosis or pulmonary embolism. N Engl J Med. 1998 Apr 23;338(17):1169-73. doi: 10.1056/NEJM199804233381701. PMID 9554856
- [Background] Buller HR, Davidson BL, Decousus H, Gallus A, Gent M, Piovella F, Prins MH, Raskob G, van den Berg-Segers AE, Cariou R, Leeuwenkamp O, Lensing AW; Matisse Investigators. Subcutaneous fondaparinux versus intravenous unfractionated heparin in the initial treatment of pulmonary embolism. N Engl J Med. 2003 Oct 30;349(18):1695-702. doi: 10.1056/NEJMoa035451. PMID 14585937
- [Background] Baron JA, Gridley G, Weiderpass E, Nyren O, Linet M. Venous thromboembolism and cancer. Lancet. 1998 Apr 11;351(9109):1077-80. doi: 10.1016/S0140-6736(97)10018-6. PMID 9660575
- [Background] Beckers MM, Verzijlbergen JF, van Buul MM, Prins MH, Biesma DH. The potential role of positron emission tomography in the detection of occult cancer in 25 patients with venous thromboembolism. Ann Oncol. 2008 Jun;19(6):1203-4. doi: 10.1093/annonc/mdn156. Epub 2008 Apr 2. No abstract available. PMID 18385199